CLINICAL TRIAL: NCT07185022
Title: a Multicenter Prospective Randomized Controlled Trial of Intra-artErial thrombolysiS for aCUte Ischemic strokE With Medium Vessel Occlusion (RESCUE MeVO)
Brief Title: Intra-arterial Thrombolysis for Acute Ischemic Stroke With Medium Vessel Occlusion
Acronym: RESCUE MeVO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Qi Li, Professor, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YX2025-105(F1)
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Cerebrovascular Disorders; Brain Diseases; Nervous System Diseases; Vascular Diseases; Ischemic Stroke; Infarction; Medium Vessel Occlusion
Keywords: Ischemic stroke; Medium vessel occlusion; Stroke; Intra-arterial thrombolysis
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Brain Diseases; Nervous System Diseases; Vascular Diseases; Ischemic Stroke; Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-arterial Thrombolysis plus Best Medical Treatment (Experimental): Patients in this group will receive intra-arterial thrombolysis plus best medical treatment.
  Interventions: Procedure: Intra-arterial Thrombolysis; Drug: Best Medical Treatment
- Best Medical Treatment (Other): Patients in this group will receive standard medical therapy in accordance with the guideline-directed management for acute ischemic stroke.
  Interventions: Drug: Best Medical Treatment

INTERVENTIONS:
Procedure: Intra-arterial Thrombolysis — rhTNK-tPA（Tenecteplase）dose: 0.4 - 0.8 mg/min, maximum dose: 16mg.
  Arms: Intra-arterial Thrombolysis plus Best Medical Treatment
Drug: Best Medical Treatment — Patients in this group will receive standard medical therapy in accordance with the guideline-directed management for acute ischemic stroke.

SUMMARY:
Acute ischemic stroke (AIS) due to medium vessel occlusion (MeVO) poses a significant clinical challenge. Recent large randomized controlled trials, DISTAL and ESCAPE-MeVO, demonstrated no significant benefit of endovascular therapy in patients with MeVO. Although intra-arterial thrombolysis has shown promise in clinical experience, robust evidence supporting its efficacy in MeVO-related AIS is still absent. To fill this gap, the RESCUE MeVO trial has been designed as a multicenter, prospective, randomized, open-label, blinded end-point (PROBE) study to evaluate the efficacy and safety of intra-arterial thrombolysis in patients with AIS caused by MeVO.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized, open-label, blinded end-point (PROBE) trial. Eligible participants will be adults (age >18 years) presenting with acute ischemic stroke (AIS) due to medium vessel occlusion (MeVO). Participants who meet all inclusion criteria and none of the exclusion criteria will be randomly assigned in a 1:1 ratio to one of two treatment arms. The control group will receive best medical management alone, while the intervention group will receive best medical management in combination with intra-arterial thrombolysis. Intra-arterial thrombolysis is performed by infusing rhTNK-tPA (Tenecteplase) proximal to the occlusion for 5-30 minutes, with the decision to continue beyond the first 5 minutes being guided by intraprocedural DSA. The primary objective of this study is to evaluate the efficacy and safety of intra-arterial thrombolysis in patients with acute ischemic stroke caused by medium vessel occlusion (MeVO). The primary endpoint is excellent outcome at 90 days, defined as a score of 0-1 on the modified Rankin Scale (mRS).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Primary medium vessel occlusion (MeVO) was detected on CTA, MRA, or DSA, involving arterial segments including M2-M3 of the middle cerebral artery (MCA), A1-A2 of the anterior cerebral artery (ACA), P1-P2 of the posterior cerebral artery (PCA), and the anterior inferior cerebellar artery (AICA), posterior inferior cerebellar artery (PICA), and superior cerebellar artery (SCA)
* The clinical symptoms were consistent with MeVO, with a NIHSS score 5 - 25, or an NIHSS score of 3-4 in the presence of disabling neurological deficits (e.g., hemianopia, aphasia, or motor dysfunction)
* Intra-arterial thrombolysis was administered within the following time windows:

  1. Acute ischemic stroke within 24 hours of symptom onset or last known well, including stroke with known onset, wake-up stroke and stroke with unknown onset;
  2. Acute ischemic stroke within 24-72 hours of onset, meeting at least one of the following imaging criteria: a.CT or MR perfusion imaging demonstrating target mismatch, defined as an ischemic core volume <30 mL, a mismatch ratio ≥1.2, and a mismatch volume ≥10 mL.; b.MRI demonstrating DWI-FLAIR mismatch, defined as the presence of acute ischemic lesions on diffusion-weighted imaging (DWI) with no corresponding hyperintense signal on FLAIR, or with FLAIR hyperintense lesions occupying less than one-third of the DWI lesion volume.
* Signed informed consent obtained

Exclusion Criteria:

* Pre-stroke mRS ≥ 2
* Secondary MeVO caused by endovascular therapy
* Neuroimaging demonstrated intracranial hemorrhage, subarachnoid hemorrhage, or other hemorrhagic disorders
* Non-contrast CT demonstrating a clearly hypodense lesion corresponding to the vascular territory
* Platelet count <100 × 10⁹/L, known bleeding tendency or coagulation factor deficiency, or oral anticoagulant therapy with an international normalized ratio (INR) >3.0
* Persistent and uncontrolled hypertension, defined as systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg
* History of intracranial hemorrhage within the past 3 months, including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, epidural hemorrhage, or subdural hemorrhage
* Presence of arteriovenous malformations or brain tumors with mass effect
* Gastrointestinal or urinary tract bleeding, or major surgery within the past 3 months
* Chronic dialysis or severe renal impairment, defined as a glomerular filtration rate (GFR) <30 mL/min or serum creatinine >220 μmol/L (2.5 mg/dL)
* Patients with known allergy to thrombolytic agents or their excipients
* Patients with known allergy to iodinated contrast agents or other established contraindications
* Pregnant or current breastfeeding
* Presence of severe systemic comorbidities with a life expectancy of less than 3 months
* Deemed unsuitable for participation by the investigator for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-02-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Excellent outcome | Time Frame: 90 ± 7 days
  Number of participants achieving an excellent outcome, defined as a modified Rankin Scale (mRS) score of 0-1 at 90 ± 7 days follow-up. The mRS is a widely used 6-point scale for assessing disability and functional outcomes after stroke, where higher scores represent worse outcomes.

SECONDARY OUTCOMES:
Ordinal distribution of mRS | 90 ± 7 days
  Ordinal distribution of the modified Rankin Scale (mRS) at 90 ± 7 days. The mRS is a widely used 6-point scale for assessing disability and functional outcomes after stroke, where higher scores represent worse outcomes.
Functional independence | Frame: 90 ± 7 days
  The proportion of patients achieving functional independence, defined as a modified Rankin Scale (mRS) score of 0-2 at 90 ± 7 days follow-up. The mRS is a widely used 6-point scale for assessing disability and functional outcomes after stroke, where higher scores represent worse outcomes.
Poor functional outcome | 90 ± 7 days
  Number of participants achieving a poor functional outcome, defined as a modified Rankin Scale (mRS) score of 4-6 at 90 ± 7 days follow-up. The mRS is a widely used 6-point scale for assessing disability and functional outcomes after stroke, where higher scores represent worse outcomes.
Early neurological deterioration | 24 ± 12 hours
  The proportion of patients with an increase of ≥ 4 points in the National Institutes of Health Stroke Scale (NIHSS) score, within 24 ± 12 hours post-randomization. The NIHSS is a standardized 11-item assessment tool designed to quantify neurological deficits in patients with acute stroke. The total score ranges from 0 to 42, with higher values indicating more severe deficits.
Any neurological improvement | 24 ± 12 hours
  The proportion of patients with a reduction of ≥ 2 points in the National Institutes of Health Stroke Scale (NIHSS) score from baseline at 24 ± 12 hours post-randomization. The NIHSS is a standardized 11-item assessment tool designed to quantify neurological deficits in patients with acute stroke. The total score ranges from 0 to 42, with higher values indicating more severe deficits.
Early neurological improvement | 24 ± 12 hours
  The proportion of patients with a reduction of ≥ 4 points in the National Institutes of Health Stroke Scale (NIHSS) score from baseline at 24 ± 12 hours post-randomization. The NIHSS is a standardized 11-item assessment tool designed to quantify neurological deficits in patients with acute stroke. The total score ranges from 0 to 42, with higher values indicating more severe deficits.

OTHER OUTCOMES:
Symptomatic intracranial hemorrhage | 24 ± 12 hours
  The incidence of symptomatic intracranial hemorrhage within 24 ± 12 hours post-randomization
All cause mortality | 90 ± 7 days
  All cause mortality at 90 ± 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Li, professor, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second (Affiliated) Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided